CLINICAL TRIAL: NCT00749034
Title: Phase I Open Label, Randomized, Controlled, Dose-Escalation Study to Evaluate Safety and Immunogenicity of VPM1002 in Comparison With BCG in Healthy Male Volunteers Stratified for History of BCG-Vaccination
Brief Title: Dose-Escalation Study on Safety and Immunogenicity of VPM1002 in Comparison With BCG in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Responsible Party: Dr. Hans-Heinrich Henneicke - v. Zepelin / CPM, Vakzine Projekt Management GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VPM1002-GE-1.01TB
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-04

CONDITIONS: Tuberculosis; Healthy
Keywords: Safety; Immunogenicity; Tuberculosis; Vaccination; Vaccination against tuberculosis; Safety and immunogenicity of VPM1002 in comparison with BCG
MeSH Terms: conditions — Tuberculosis | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): VPM1002 in three dosages
  Interventions: Biological: VPM1002
- 2 (Active Comparator): BCG
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: VPM1002 — live vaccine
  Arms: 1
Biological: BCG — commercially available live vaccine BCG
  Arms: 2

SUMMARY:
Goal of VPM is the development of a recombinant urease C-deficient listeriolysin expressing BCG vaccine strain (VPM1002) as a safe, well tolerated and efficacious vaccine against TB for residents in endemic areas and persons at risk in non-endemic areas. The new live vaccine VPM1002 should be at least as potent as the currently used BCG vaccine and should cause fewer side effects (Kaufmann, 2007; Grode et al., 2005). It is formulated as lyophilised bacteria to be resuspended before intradermal injection. First application of VPM1002 in human male volunteers will evaluate its safety, local and systemic tolerability as well as its immunogenicity. The study has a dose-escalating sequential design with comparison to commercially available BCG. 80 volunteers in Germany will randomly be allocated to 4 groups each with 20 volunteers stratified for their history of BCG-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers 18 to 55 years of age.
2. Healthy (medical history, physical examination, vital signs, ECG and laboratory tests at screening).
3. No signs of active or latent tuberculosis infection.
4. BMI of 19 - 30 kg/m2.
5. Subjects must be able and willing to comply with the study protocol, available and willing to complete all study measurements and have signed an Informed Consent form approved by the Ethics Committee.
6. Intention not to travel to endemic regions for tuberculosis (such as Africa, Asia, former USSR) and reachable by phone during the whole study period (6 months).
7. Negative test for HIV1 and HIV2, hepatitis B surface antigen and antibody to hepatitis C virus .
8. No anamnestic evidence for a primary or secondary immunodeficiency.
9. No skin eczema lesion at the intended injection site.
10. No anamnestic predisposition for scarring badly or for keloid formation.
11. No other vaccination during eight weeks before and during the follow-up period of the current study. If a vaccination is necessary during this period, the volunteer will be withdrawn from the study.
12. No participation in another clinical trial within 3 months before study vaccination and the 6 months of the current study.
13. Able and willing to abstain from physical exercise 24 hours before screening examination, and from 24 hours before admission until discharge from the clinic.
14. No blood donation for non study-related purposes during the entire duration of the study.
15. normal sonographic liver imaging

Exclusion Criteria:

For the group of volunteers who were vaccinated with a BCG vaccine:

â€¢ Tuberculin-PPD-in-vivo-test equal or more than 10 mm at baseline

For the group of naive volunteers:

â€¢ Tuberculin-PPD-in-vivo-Test equal or more than 1 mm at baseline

For all volunteers

1. systemic disorders which could interfere with the interpretation of the study results or compromise the health of the volunteers.
2. BCG-vaccination during 10 years before study vaccination.
3. Acute fever or fever in the last 7 days before dosing.
4. Any malignant condition.
5. Concomitant treatment with medication that may affect immune function during 3 months before study vaccination and the 6 months of current study.
6. Treatment with blood products or Immunoglobulins in the past 6 months up to end of study.
7. Any clinically significant laboratory abnormalities on screened blood samples.
8. A history of drug or alcohol abuse.
9. History of anaphylaxis or severe allergic reactions.
10. Positive test for drugs of abuse on urine testing at screening or admission.
11. Known allergies to any component of the investigational or reference product or known history of severe skin reaction against the Tuberculin test.
12. Professional or regular contact with life animals for food production.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety: physical examination, vital signs, ECG, liver sonography, chest X-ray, laboratory safety parameters (including haematology, coagulation, clinical chemistry and urinalysis), tolerability, recording of concomitant medication and adverse events | days -1, 1, 2, 3, 5, 11, 29, 57 and month 6

SECONDARY OUTCOMES:
Immunogenicity: LST for PPD with subsequent IFN-gamma specific ELISA on supernatants of PBMC | baseline, days 29, 57, month 6
Immunogenicity: ELISPOT for the number of IFN-gamma secreting PBMC after stimulation with PPD | baseline, days 29, 57, month 6
Immunogenicity: whole blood stimulated with PPD and measuring IFN-gamma in the plasma by ELISA | baseline, days 29, 57, month 6
ICS for IFN-gamma, TNF-alpha and IL-2 in CD4+ and CD8+ lymphocytes upon stimulation with PPD | baseline, days 29, 57 and month 6
Immunogenicity: ICS with other triple combinations of markers in CD4+ and CD8+ lymphocytes upon stimulation with PPD | baseline, days 29, 57 and month 6
Immunogenicity: TB85B as recall antigen for ELISA, ELISPOT, WBA and ICS | baseline, days 29, 57 and month 6
Immunogenicity: serum antibodies against PPD or AG85B | baseline, days 29, 57 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schrödter, MD, Principal Investigator — FOCUS CDD GmbH
Locations (1):
- Focus Clinical Drug Development GmbH, Neuss, Germany

REFERENCES:
- [Derived] Choi SW, Han S, Shim WJ, Choi DJ, Kim YJ, Yoo BS, Hwang KK, Jeon HK, Shin MS, Ryu KH. Impact of Heart Rate Reduction with Maximal Tolerable Dose of Bisoprolol on Left Ventricular Reverse Remodeling. J Korean Med Sci. 2018 May 11;33(25):e171. doi: 10.3346/jkms.2018.33.e171. eCollection 2018 Jun 18. PMID 29915522
- [Derived] Grode L, Ganoza CA, Brohm C, Weiner J 3rd, Eisele B, Kaufmann SH. Safety and immunogenicity of the recombinant BCG vaccine VPM1002 in a phase 1 open-label randomized clinical trial. Vaccine. 2013 Feb 18;31(9):1340-8. doi: 10.1016/j.vaccine.2012.12.053. Epub 2013 Jan 3. PMID 23290835
- See also: Background Information on VPM1002 — http://www.vakzine-manager.de/index.php?id=169&L=1